CLINICAL TRIAL: NCT03434366
Title: Intranasal Ketamine With Dexmedetomidine for the Treatment of Children With Autism Spectrum Disorder
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: The effects are not good
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Ying Jun She, MD, Department of Anesthesiology, Guangzhou Women and Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: intranasal ketamine
Record Dates: First submitted 2018-01-28; First posted 2018-02-15 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; ketamine; dexmedetomidine
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Ketamine; Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ketamine and dexmedetomidine group (Experimental): intranasal ketamine and dexmedetomidine was treated in the children
  Interventions: Drug: ketamine and dexmedetomidine
- ketamine group (Experimental): intranasal ketamine was treated in the children
  Interventions: Drug: ketamine
- control group (Placebo Comparator): intranasal insaline was used in the children
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: ketamine and dexmedetomidine — intranasal ketamine and dexmedetomidine for treatment for autism spectrum disorder
  Other Names: intranasal ketamine and dexmedetomidine
  Arms: ketamine and dexmedetomidine group
Drug: ketamine — intranasal ketamine for treatment for autism spectrum disorder
  Other Names: intranasal ketamine
  Arms: ketamine group
Drug: Saline — intranasal saline for treatment for autism spectrum disorder
  Other Names: intranasal saline
  Arms: control group

SUMMARY:
Autism spectrum disorder (ASD) is a life-long neurodevelopmental disorder characterized by qualitative abnormalities in reciprocal social interactions and patterns of communication, and by a restricted, stereotyped, repetitive repertoire of interests and activities. The use of medications in adolescents and young adults with ASD is extremely common. However, few data address the effectiveness and harms of medications specifically in this population.

The purpose of the study is to determine the efficacy and safety of intranasal ketamine with dexmedetomidine in children with ASD.

DETAILED DESCRIPTION:
The use of medications in adolescents and young adults with ASD is extremely common. few data address the effectiveness and harms of medications specifically in this population. A previous study reported the first case study demonstrating clinical improvement in mood and eye fixation scores from intranasal ketamine treatment in a "complicated" subject with autism spectrum disorderHowever,The purpose of the study is to determine the efficacy and safety of intranasal ketamine with dexmedetomidine in children with ASD.

ELIGIBILITY:
Inclusion Criteria:

1. meet autism diagnostic criteria based on DSM-5/ADI-R/ADOS
2. children aged 2 years through 15 years of age
3. parents/guardians can cooperate with the study and sign informed consent
4. ASA score I or II

Exclusion Criteria:

1. with epilepsy or other genetic diseases
2. changes in drugs or in any intervention during the study
3. Presence of cardiac disease including coronary artery disease, congestive heart failure, or uncontrolled hypertension per medical history
4. Airway instability, tracheal surgery, or tracheal stenosis per medical history.
5. History of drug or alcohol abuse
6. Central nervous system masses or hydrocephalus per medical history

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2018-01-20 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Autism Diagnostic Interview Revised (ADI-R) | change from baseline at 2, 5 and 12 weeks
  The Autism Diagnostic Interview Revised is an investigator-based semi-structured diagnostic interview, The ADI-R provides empirically derived diagnostic algorithms for three subdomains of qualitative impairments. The social interaction domain includes questions about emotional sharing, offering and seeking comfort, social smiling, and social responding comprising four subscores. The second domain (communication) assesses stereotyped expressions, pronoun reversal, and the social usage of language (B1-B4). In the third domain repetitive and stereotyped behavior as hand- and finger mannerisms, unusual sensory interest or activities are investigated by four subscales. Most items are scored from zero to three, relying on the interviewer to make judgements on child's behaviour based on the recall of information from parents/carers. . A total score is then calculated for each of the three subdomains. The ADI-R has an algorithm for autism based on scores in these three areas and on onset.
Autism Diagnostic Observation Schedule (ADOS) | change from baseline at 2, 5 and 12 weeks
  The Autism Diagnostic Observation Schedule (ADOS) is a semi-structured assessment of communication, social interaction and play or imaginative use of materials for individuals suspected of having autism or other ASD. It consists of four modules, each of which is appropriate for children, adolescents and adults of differing developmental and language levels, ranging from no expressive or receptive language to verbally fluent adults. The examiner selects the module that is most appropriate for a particular child, adolescent on the basis of his/her expressive language level and chronological age. Selected algorithm items relating to social interaction and communication are then entered into an algorithm. The scores must meet the separate cut-offs for both the communication and social domains and the cut-off for the summation of the two. Repetitive behaviours are recorded and coded as part of the clinical observations but do not contribute to the ADOS summary algorithm.

SECONDARY OUTCOMES:
autism behavior checklist (ABC) | change from baseline at 2, 5 and 12 weeks
  ABC is a scale used for nonadaptive behaviors created to screen and indicate the probability of a diagnosis of autism. The questionnaire approaches 57 atypical behaviors related to five areas: sensorial, relational, use of body and objects, and social skills. Scales> 67 was diagnosised ASD, compare the change in scales in different time point(from baseline to endpoint)
magnetic resonance spectroscopy(MRS) | change from baseline at 5 and 12 weeks
  compare the metabolite concentrations and ratios in brain from Baseline to Endpoint (NAA,Glu,Gln,Cho,Cr,mI)
Childhood Autism Rating Scale (CARS) | change from baseline at 2, 5 and 12 weeks
  CARS assesses the child on a scale from 1 to 4 in each of 15 dimensions or symptoms (including the ability to relate to people, emotional response, imitation, body use, object use, listening response, fear or nervousness, verbal communication, nonverbal communication, activity level, level and reliability of intellectual response, adaptation to changes, visual response, taste, smell and touch responses and general impressions). A total score of at least 30 strongly suggests the presence of autism. Children who score between 30 and 36 have mild-to-moderate autism while those with scores between 37 and 60 have severe autism. Change in CARS from Baseline to Endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Zhao, Doctor, Principal Investigator — Guangzhou Women and Children's Medical Center
Locations (1):
- Guangzhou Women and Children Medical Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided